CLINICAL TRIAL: NCT05338099
Title: Open-label, Dose-escalation, Phase 1 Clinical Trial to Determine the Safety and Dose of EN001 in Patients With Duchenne Muscular Dystrophy(DMD)
Brief Title: Determine the Safety and Dose of EN001 in Patients With Duchenne Muscular Dystrophy(DMD)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ENCell (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ENCell_2020_01
Record Dates: First submitted 2022-01-06; First posted 2022-04-20 (Actual); Last update posted 2024-08-30 (Actual); Status verified 2024-08

CONDITIONS: Duchenne Muscular Dystrophy
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dose group A (Low dose) (Experimental): Participants will receive EN001 intravenously (IV) once on Day 1. Before 30 minutes EN001 dosing, there will be premedication (solu-cortef 1-2 mg/kg + Lorazepam 0.1 mg/kg (max 2 mg) + Ondansetron (5 mg/m^2) + Chlorpheniramine (1 mg for 2~6 years old; 2 mg for 6~12 years old; 4 mg for over 12 years old)+ Acetaminophen) administered to assure safety of participants from issues such as immune rejection, due to the process of thawing in a frozen state of EN001.
  Interventions: Drug: EN001
- Dose group B (High dose) (Experimental): Participants will receive EN001 intravenously (IV) once on Day 1. Before 30 minutes EN001 dosing, there will be premedication (solu-cortef 1-2 mg/kg + Lorazepam 0.1 mg/kg (max 2 mg) + Ondansetron (5 mg/m^2) + Chlorpheniramine (1 mg for 2~6 years old; 2 mg for 6~12 years old; 4 mg for over 12 years old)+ Acetaminophen) administered to assure safety of participants from issues such as immune rejection, due to the process of thawing in a frozen state of EN001.
  Interventions: Drug: EN001

INTERVENTIONS:
Drug: EN001 — EN001 intravenously (IV) in the treatment of Duchenne Muscular Dystrophy (DMD) Dosage for each group is as follows.
  Dose group A (Low dose): 5.0x10^5 cells/kg
  Other Names: EN001 (Allogeneic early-passage Wharton's jelly-derived mesenchymal stem cells)
  Arms: Dose group A (Low dose)
Drug: EN001 — EN001 intravenously (IV) in the treatment of Duchenne Muscular Dystrophy (DMD) Dosage for each group is as follows.
  Dose group B (High dose): 2.5x10^6 cells/kg
  Other Names: EN001 (Allogeneic early-passage Wharton's jelly-derived mesenchymal stem cells)
  Arms: Dose group B (High dose)

SUMMARY:
Open-label, Dose-escalation, Phase 1 Clinical Trial to Determine the Safety and Dose of EN001 in Patients with Duchenne Muscular Dystrophy(DMD)

DETAILED DESCRIPTION:
It is the first in human (FIH), 3+3 design clinical trial to evaluate the safety and tolerability and determine the maximum tolerated dose (MTD) of EN001 (allogeneic umbilical cord-derived mesenchymal stem cells) in the treatment of Duchenne Muscular Dystrophy (DMD).

ELIGIBILITY:
Inclusion Criteria:

1. Those aged 2 to 18 years old
2. Male
3. Those who are diagnosed with DMD due to a mutation in the dystrophin gene identified by a genetic test
4. Phenotypic evidence of DMD

   * Clinical signs or symptoms (proximal weakness, waddling gait, Gowers maneuver)
   * Elevated serum creatine kinase level
5. Those who have been using systemic corticosteroids at a stable dose for 24 weeks prior to screening and are expected to maintain the constant dose throughout the study period
6. Those who agree to use effective contraceptive measures until the short-term follow-up period of the clinical trial. In addition, their partner must also use a medically acceptable method of contraception (ie, oral contraceptives for women) for the same period.
7. Those who are willing to agree with the ICF and whose parent or representative is willing to provide written consent for the subject's participation in the clinical trial

Exclusion Criteria:

1. Those who have clinical signs or symptoms of cardiomyopathy, defined as LVEF <50% on echocardiography at screening
2. If ventilatory support is required during the day or if invasive mechanical ventilation via tracheostomy is used (Non-invasive ventilation such as positive pressure ventilation is allowed at night)
3. If hepatitis B core antibody and hepatitis C antibody are positive
4. If there is a history of major surgery within 12 weeks or it is expected during the study period
5. Those who have been exposed to gene therapy or genome editing within 24 weeks from the screening
6. Those who have experience with stem cell therapy
7. Those who have been administered Translarna granules (Ataluren) within 24 weeks from the screening
8. Those who are receiving treatment (other than corticosteroids) that may affect muscle strength or function within 12 weeks prior to screening
9. If laboratory test values are abnormal at the time of screening

   * Hemoglobin <10 g/dL
   * Serum albumin <2.5 g/dL
   * Platelet count <50,000/ml
   * Abnormal GGT or total bilirubin (>laboratory's upper limit of normal)
   * Abnormal renal function (Serum creatinine >1.5 Times laboratory's upper limit of normal)"
10. Those with significant neuromuscular or genetic diseases other than DMD
11. Those with significant heart, lung, liver, kidney, hematological, immunological, behavioral disease, or other clinically significant diseases including malignant tumors
12. Those who have a previous or current medical condition that may adversely affect the safety of the subject, make it difficult to complete treatment, or affect the evaluation of clinical trial results at the discretion of the investigator
13. Those who do not have the will or ability to comply with clinical trial procedures at the discretion of the investigator

Ages: 2 Years to 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 7 (Actual)
Dates: Start 2022-01-18 (Actual); Primary Completion 2022-12-28 (Actual); Study Completion 2022-12-28 (Actual)

PRIMARY OUTCOMES:
Number of participants of any Adverse Events (AEs)/Serious Adverse Events (SAEs) related investigational product | Week 12 after treatment
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0
Determination of Dose-limiting toxicity (DLT) levels of EN001 | Up to Week 2 after dosing on Day 0
  Among the adverse events occurring for 2 weeks after administration of the investigational product, Grade 3 or higher adverse events according to CTCAE 5.0
Determination of Maximum tolerated dose (MTD) levels of EN001 | Up to Week 2 after dosing on Day 0
  Among the adverse events occurring for 2 weeks after administration of the investigational product, Grade 3 or higher adverse events according to CTCAE 5.0 Maximum tolerated dose defines the evaluated maximum dose level in which greater than two participants of six participants experience Dose-limiting toxicity (DLT) under the dose level. The dose level where two participants of six participants experience DLT will be the maximum tolerated dose.
Number of participants with Vital Signs abnormalities | Week 12 after screening
  Vital Signs include blood pressure (mmHg), pulse (times/minute), respiratory rate (times/minute), and body temperature (℃) and will be assessed by CTCAE v 5.0 to evaluate safety and tolerability of EN001.
  The number of participants with at least one potentially clinically significant abnormal vital sign finding were reported as treatment emergent adverse events (TEAEs).
Number of participants with clinically significant abnormalities of Physical Examinations | From screening up to Week 12
  Physical Examinations include general appearance, head, ears/eyes/nose/throat, cardiovascular, respiratory, abdomen, skin, lymph nodes, extremities, musculoskeletal and neurologic and will be assessed by CTCAE v 5.0 to evaluate safety and tolerability of EN001.
  Number of participants with potentially clinically significant abnormalities in physical examinations were reported as TEAEs.
Number of participants with abnormalities of Laboratory Parameters | From screening up to Week 12
  Laboratory Parameters include hematology, chemistry laboratory tests, urinalysis, coagulation test and plasma viral load test and will be assessed by CTCAE 5.0 to evaluate safety and tolerability of EN001.
  Number of participants with at least one potentially clinically significant abnormal finding were reported as TEAEs.
Number of participants with abnormalities of 12-lead Electrocardiography (ECG) | From screening to baseline on Day 0 (Predose to end of infusion and 90 min after completion of infusion)
  Categorical summarization ECG criteria were as follows:
  1. QT interval, QTcB, QTcF and QTcP: increase from baseline >30 millisecond [ms] or 60 ms; absolute value > 450 ms, >480 ms, and > 500 ms;
  2. heart rate (HR): change from baseline ≥20 beats per minute [bpm] and absolute value≤50 bpm or ≥120 bpm;
  3. PR interval: absolute value ≥220 ms and increase from baseline≥20 ms;
  4. QRS: ≥120 ms.

SECONDARY OUTCOMES:
Incidence of adverse events (AEs) | From screening to the end of treatment/withdrawal visit (up to approximately 5 years per subject)
  Occurrence of any adverse reactions, development of new blood clots, tumors, immune responses (like autoimmune reactions) and death, and/or serious adverse events related investigational product will be summarized by actual treatment groups respectively.
Number of participants with abnormalities of Vital Signs, Physical Findings, and Laboratory Parameters | From screening to the end of treatment/withdrawal visit (up to approximately 5 years per subject)
  Abnormalities of Vital Signs, Physical Findings, and Laboratory parameters (as described above) will be collected and analyzed, and then assessed by CTCAE 5.0 to evaluate the long-term safety of EN001.
Rate of change at the time of visit compared to baseline (percent [%]) in CK level | From screening up to the end of support (up to approximately 5 years per subject at each visit)
  Creatinine kinase (CK) level will be collected and analyzed to evaluate the exploratory efficacy of EN001.
  - CK level(%) = (CK level after dosing - CK level in baseline)/(CK level in baseline)*100
Change from baseline in Function tests | Screening and baseline on Day -1 (up to approximately 5 years per subject after Week 12)
  Function tests measured by North Star Ambulatory Assessment (NSAA), Six Minute Walk Test (6MWT), Myometry. and Lung capacity (and only K-Cross Motor Function Measure (KGMFM) will be performed under 5 years old) will be collected and analyzed to evaluate the exploratory efficacy of EN001.
  - Function tests = value in visit - value in baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea